CLINICAL TRIAL: NCT03693781
Title: Colchicine for Amyotrophic Lateral Sclerosis: a Phase II, Randomized, Double Blind, Placebo Controlled, Multicenter Clinical Trial
Brief Title: Colchicine for Amyotrophic Lateral Sclerosis
Acronym: Co-ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Collaborators: University of Modena and Reggio Emilia (Other); University of Turin, Italy (Other); Istituto Auxologico Italiano (Other); IRCCS National Neurological Institute "C. Mondino" Foundation (Other); University of Bari (Other); IRCCS San Raffaele (Other); University of Padova (Other); University of Milan (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other); University of Campania Luigi Vanvitelli (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, JESSICA MANDRIOLI, Principal Investigator, Azienda Ospedaliero-Universitaria di Modena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Co-ALS
Record Dates: First submitted 2018-09-30; First posted 2018-10-03 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; stress granules; HSPB8; protein quality control; colchicine; ALSFRS-r; survival; safety
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Three arms of 18 patients each; in two arms two colchicine dosages will be tested compared to placebo in the control arm. The three arms will undergo treatment vs placebo in parallel
Who Masked: Participant, Investigator
Masking Description: placebo will be unrecognizable from active treatment (both in tablets)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Colchicine 0.01mg/kg/day + Riluzole 100 mg (Active Comparator): Oral colchicine will be administered at fast, at specified dose pro kilograms for 30 weeks, while taking Riluzole 100 mg/day
  Interventions: Drug: Colchicine 1 MG Oral Tablet
- Colchicine 0.005 mg/kg/day + Riluzole 100 mg (Active Comparator): Oral colchicine will be administered at fast, at specified dose pro kilograms for 30 weeks, while taking Riluzole 100 mg/day
  Interventions: Drug: Colchicine 1 MG Oral Tablet
- Placebo + Riluzole 100 mg (Placebo Comparator): Placebo pills will be administered at fast, while taking Riluzole 100 mg/day
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Colchicine 1 MG Oral Tablet — Colchicine tablets depending on arm (0.01 mg/kg/day, 0.005 mg/kg/day, placebo) and on weight (>70 kg or <71 kg) for 30 weeks of duration.
  Arms: Colchicine 0.01mg/kg/day + Riluzole 100 mg
Drug: Colchicine 1 MG Oral Tablet — Colchicine tablets depending on arm (0.01 mg/kg/day, 0.005 mg/kg/day, placebo) and on weight (>70 kg or <71 kg) for 30 weeks of duration.
  Arms: Colchicine 0.005 mg/kg/day + Riluzole 100 mg
Drug: Placebo Oral Tablet — Corresponding tablets for 30 weeks
  Arms: Placebo + Riluzole 100 mg

SUMMARY:
The study evaluates the effects of two different Colchicine doses (0.01mg/kg/day or 0.005 mg/kg/day) compared to placebo in Amyotrophic Lateral Sclerosis (ALS) patients. Disease progression as defined by changes in ALSFRS-r is the primary outcome measure. Other measures of clinical progression and survival, together with safety and tolerability of Colchicine in ALS patients will be assessed.

DETAILED DESCRIPTION:
Recent evidence supports the disruption of the ubiquitin-proteasome-system and autophagy as central events in ALS. ALS is characterized by the presence of misfolded proteins prone to oligomerize into aggregates, which exert a toxic effect by affecting several intracellular functions. Heat shock protein B8 (HSPB8) recognizes and promotes the autophagy-mediated removal of misfolded mutant SOD1 and TDP-43 fragments from ALS motor neurons (MNs). Moreover, HSPB8-BAG3-HSP70 maintains the so called "granulostasis", a surveillance mechanism that avoids the conversion of dynamic stress granules (SGs) into aggregation-prone assemblies, which are a hallmark of ALS.

Colchicine enhances the expression of HSPB8 and of several autophagy players while blocking TDP-43 accumulation in neurons. Moreover, given the cross-talk between infalmmation and autophagy, the well-known antinflammatory action of Cochicine may contribute to cell homeostasis.

Based on these premises, this is a phase II randomized, double-blind, placebo-controlled, multicenter (9 MND Centres in Italy: 2 centres in Milan, Pavia, Turin, Modena, Padua, Rome, Naples, Bari), clinical trial to test efficacy of Colchicine in ALS.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a laboratory supported, clinically "probable" or "definite" amyotrophic lateral sclerosis according to the Revised El Escorial criteria (Brooks, 2000)
* Sporadic ALS
* ALS phenotypes: classic or bulbar
* Female or male patients aged between 18 and 80 years old
* Disease duration from symptoms onset no longer than 18 months at the screening visit
* Patients treated with a stable dose of Riluzole (100 mg/day) for at least 30 days prior to screening
* Patients with a weight > 50 kg and a BMI ≥18
* Patients with a FVC (Forced Vital Capacity) equal or more than 65 % predicted normal value for gender, height, and age at the screening visit Patients able and willing to comply with study procedures as per protocol
* Patients able to understand, and capable of providing informed consent at screening visit prior to any protocol-specific procedures
* Use of highly effective contraception

Exclusion Criteria:

* Prior use of Colchicine
* Prior allergy/sensitivity to Colchicine
* Receiving Colchicine or other anti-inflammatory drugs (such as corticosteroids, methotrexate, anti-neoplastic, Interleukin 1-1b antagonist, Tumor necrosis factor-alpha inhibitor)
* Receiving food or co-medications such as strong-moderate cytochrome P450 3A4 inhibitors that will result in elevated plasma level of Colchicine
* Inflammatory disorders (SLE, Rheumatoid arthritis, connective tissue disorder) or chronic infections (HIV, hepatitis B or C infection) or significant history of malignancy
* Severe renal (eGFR< 30ml/min/1.73m2), or liver failure or liver aminotransferase (ALT/AST > 2x Upper limit of normal),
* Existing blood dyscrasia (e.g., myelodysplasia)
* White blood cells<4,000/mm³, platelets count<100,000/mm³, hematocrit<30%
* Severe comorbidities (heart, renal, liver failure), autoimmune diseases or any type of interstitial lung disease
* Patients who underwent non invasive ventilation, tracheotomy and /or gastrostomy
* Women who are pregnant or breastfeeding
* Participation in pharmacological studies within the last 30 days before screening
* Patients with the following ALS phenotypes: flail arm, flail leg, UMN-p, respiratory, PLS, progressive muscular atrophy.
* Patients with familial ALS defined as presence of at least one first degree family member (parents/son/daughter/brother/sister) affected by ALS.
* Patients with known pathogenic mutations (SOD1, TARDBP, FUS, C9ORF72).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Decrease in ALS disease progression as measured by ALS Functional rating Scale Revised (ALSFRS-R) | comparison between baseline and treatment end (week 30)
  ALSFRS-R is a scale that measures disability in ALS; the scores range from 0 (maximum disability, the worst score) to 48 (no disability, the best score). We will measure total score changes from baseline to week 30 in treatment and placebo arms.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (safety and tolerability) | week 30 and 54
  Number of serious adverse events (SAEs) and AEs in placebo and treatment arms
Tracheostomy-free survival rate | Up to week 54
  Overall survival from randomization to date of death or tracheostomy
Changes in Forced Vital Capacity (FVC) | Up to week 54
  Changes in FVC score from baseline to week 8, 18, 30, 54 in treatment and placebo arms.
Changes in quality of life | at 8,18,30 and 54 week
  Changes in Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) from baseline to week 8, 18, 30 and week 54, in placebo and treatment arms
enhancement of autophagy | at week 30 and 54, compared to baseline
  assessment of mRNA and protein levels of p62, LC3, TFEB, ATGs, HSPB8, BAG3, BAG1, HSP70, and HSF1, in patients' PBMCs, lymphoblasts and fibroblasts (transcriptome profile);
changes in stress granules size, number and composition | at week 30 compared to baseline
  identification of changes in stress granules response and composition in patients' fibroblasts and lymphoblasts will be carried out by measuring granules size, number and composition by confocal microscopy using automated systems. The aberrant recruitment or sequestration of specific mRNA inside stress granules will be assessed by FISH using specific probes, followed by densitometric analysis as previously described by Gareau et al. (2011).
quantification of insoluble species | at week 30 compared to baseline
  assessment of overall levels and the relative ratio between soluble and insoluble species of TDP-43, TDP-43 fragments, SQSTM1/p62, UBQLN, OPTN in fibroblasts and lymphoblasts derived from the same patients
modifications on extracellular vesicles secretion in blood and CSF | at week 30 compared to baseline
  assessment of TDP-43, hyperphosphorylated TDP-43, SQSTM1/p62, UBQLN and OPTN in extracellular vesicles by plasma and CSF.
effects on biomarkers of neurodegeneration | at week 30 compared to baseline
  creatinine, albumin, CK, and vitamin D in plasma as markers of disease severity; phosphorylated neurofilaments heavy chain
effects on biomarkers of inflammation | at week 30 compared to baseline
  assessment of plasma/CSF IL18, its endogenous inhibitor IL-18BP, MCP1 and IL17

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Mandrioli, Principal Investigator — Azienda Ospedaliero-Universitaria di Modena
Locations (8):
- Italy (8):
  - Centro Sla, University of Bari, Bari
  - Centro Sla, Istituto Auxologico Italiano, University of Milano, Milano, Milan
  - Irccs Carlo Besta, Milan
  - Irccs St. Raffaele Institute of Milano, Milan
  - Centro Sla, Ospedale Civile S. Agostino Estense, A.O.U. Modena, Modena
  - Università della Campania Gianluigi Vanvitelli, Napoli
  - Als Centre, "C. Mondino" National Neurological Institute, University of Pavia, Pavia
  - , Neuromuscular Omnicentre Centre, Rome, Catholic University, Rome, Roma

IPD SHARING:
Plan to Share IPD: Yes
de-identified individual participant data will be made available after study completion upon specific request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available at study completion (after final data analysis)
Access Criteria: specific personal request by the subject

REFERENCES:
- [Background] Thomas M, Alegre-Abarrategui J, Wade-Martins R. RNA dysfunction and aggrephagy at the centre of an amyotrophic lateral sclerosis/frontotemporal dementia disease continuum. Brain. 2013 May;136(Pt 5):1345-60. doi: 10.1093/brain/awt030. Epub 2013 Mar 9. PMID 23474849
- [Background] Cadwell K. Crosstalk between autophagy and inflammatory signalling pathways: balancing defence and homeostasis. Nat Rev Immunol. 2016 Nov;16(11):661-675. doi: 10.1038/nri.2016.100. Epub 2016 Oct 3. PMID 27694913
- [Background] Crippa V, D'Agostino VG, Cristofani R, Rusmini P, Cicardi ME, Messi E, Loffredo R, Pancher M, Piccolella M, Galbiati M, Meroni M, Cereda C, Carra S, Provenzani A, Poletti A. Transcriptional induction of the heat shock protein B8 mediates the clearance of misfolded proteins responsible for motor neuron diseases. Sci Rep. 2016 Mar 10;6:22827. doi: 10.1038/srep22827. PMID 26961006
- [Background] Crippa V, Cicardi ME, Ramesh N, Seguin SJ, Ganassi M, Bigi I, Diacci C, Zelotti E, Baratashvili M, Gregory JM, Dobson CM, Cereda C, Pandey UB, Poletti A, Carra S. The chaperone HSPB8 reduces the accumulation of truncated TDP-43 species in cells and protects against TDP-43-mediated toxicity. Hum Mol Genet. 2016 Sep 15;25(18):3908-3924. doi: 10.1093/hmg/ddw232. Epub 2016 Jul 27. PMID 27466192
- [Background] Cristofani R, Crippa V, Vezzoli G, Rusmini P, Galbiati M, Cicardi ME, Meroni M, Ferrari V, Tedesco B, Piccolella M, Messi E, Carra S, Poletti A. The small heat shock protein B8 (HSPB8) efficiently removes aggregating species of dipeptides produced in C9ORF72-related neurodegenerative diseases. Cell Stress Chaperones. 2018 Jan;23(1):1-12. doi: 10.1007/s12192-017-0806-9. Epub 2017 Jun 12. PMID 28608264
- [Background] Cristofani R, Crippa V, Rusmini P, Cicardi ME, Meroni M, Licata NV, Sala G, Giorgetti E, Grunseich C, Galbiati M, Piccolella M, Messi E, Ferrarese C, Carra S, Poletti A. Inhibition of retrograde transport modulates misfolded protein accumulation and clearance in motoneuron diseases. Autophagy. 2017 Aug 3;13(8):1280-1303. doi: 10.1080/15548627.2017.1308985. PMID 28402699
- [Background] Carra S, Seguin SJ, Landry J. HspB8 and Bag3: a new chaperone complex targeting misfolded proteins to macroautophagy. Autophagy. 2008 Feb;4(2):237-9. doi: 10.4161/auto.5407. Epub 2007 Dec 11. PMID 18094623
- [Background] Crippa V, Sau D, Rusmini P, Boncoraglio A, Onesto E, Bolzoni E, Galbiati M, Fontana E, Marino M, Carra S, Bendotti C, De Biasi S, Poletti A. The small heat shock protein B8 (HspB8) promotes autophagic removal of misfolded proteins involved in amyotrophic lateral sclerosis (ALS). Hum Mol Genet. 2010 Sep 1;19(17):3440-56. doi: 10.1093/hmg/ddq257. Epub 2010 Jun 22. PMID 20570967
- [Background] Terkeltaub RA. Colchicine update: 2008. Semin Arthritis Rheum. 2009 Jun;38(6):411-9. doi: 10.1016/j.semarthrit.2008.08.006. Epub 2008 Oct 29. PMID 18973929
- [Background] Taylor JP, Brown RH Jr, Cleveland DW. Decoding ALS: from genes to mechanism. Nature. 2016 Nov 10;539(7628):197-206. doi: 10.1038/nature20413. PMID 27830784
- [Background] Miller RG, Mitchell JD, Moore DH. Riluzole for amyotrophic lateral sclerosis (ALS)/motor neuron disease (MND). Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD001447. doi: 10.1002/14651858.CD001447.pub3. PMID 22419278
- [Derived] Mandrioli J, Crippa V, Cereda C, Bonetto V, Zucchi E, Gessani A, Ceroni M, Chio A, D'Amico R, Monsurro MR, Riva N, Sabatelli M, Silani V, Simone IL, Soraru G, Provenzani A, D'Agostino VG, Carra S, Poletti A. Proteostasis and ALS: protocol for a phase II, randomised, double-blind, placebo-controlled, multicentre clinical trial for colchicine in ALS (Co-ALS). BMJ Open. 2019 May 30;9(5):e028486. doi: 10.1136/bmjopen-2018-028486. PMID 31152038